CLINICAL TRIAL: NCT02891499
Title: Effect of Low-level Laser Therapy on Stability and Displacement of Orthodontic Miniscrew Implants With Mediate and Immediate Force Application
Brief Title: Influence of Low-level Laser Therapy on Stability and Displacement of Orthodontic Miniscrew Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Guido Artemio Marañón Vásquez, Master of science student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: USaoPaulo-1
Record Dates: First submitted 2016-08-23; First posted 2016-09-07 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Displacement of Other Bone Devices, Implants and Grafts; Mechanical Complication of Other Bone Devices, Implants and Grafts
Keywords: Miniscrews; Mini-implants; Temporal anchorage devices; Bone screws; Stability; Displacement; Low-level laser therapy; Cone-beam computed tomography; Resonance frequency analysis; Orthodontic; Orthodontic miniscrew implant
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LLLT + immediate force (Experimental): Use of Low-level laser therapy and not mediate orthodontic force application (150 gF the day of the implantation).
  Interventions: Procedure: Low-level laser therapy
- LLLT + mediate force (Experimental): Use of Low-level laser therapy and mediate orthodontic force application (150 gF 4 weeks after the day of the implantation).
  Interventions: Procedure: Low-level laser therapy; Procedure: Mediate force application
- Immediate force application (No Intervention): Not mediate orthodontic force application (150 gF the day of the implantation), without use of Low-level laser therapy.
- Mediate force application (Experimental): Mediate orthodontic force application (150 gF 4 weeks after the day of the implantation), without use of Low-level laser therapy.
  Interventions: Procedure: Mediate force application

INTERVENTIONS:
Procedure: Low-level laser therapy — 1. Immediate post-operative period (implantation day) Red emission (660 nm) Energy density: 4 J/cm2 Power: 0.1W Irradiation area: 0,5 cm2 One application, 10 seconds of non-contact irradiation (01 point at the area surrounding the miniscrew) at a distance of 15,5 mm.
  2. Mediate post-operative period (after implantation day) Infrared emission (808 nm) Energy density: 8 J/cm2 Power: 0.1W Irradiation area: 0,5 cm2 6 applications every 48 hours after the day of implantation, 20 seconds of non-contact irradiation (01 point on the area surrounding the miniscrew) at a distance of 15,5 mm.
  Arms: LLLT + immediate force; LLLT + mediate force
Procedure: Mediate force application — Mediate force application protocol: orthodontic force application (150 gF) 4 weeks after the day of the implantation.
  Arms: LLLT + mediate force; Mediate force application

SUMMARY:
The purpose of this study is to evaluate the effect of Low level laser therapy on stability and displacement of orthodontic miniscrew implants using two different force application protocols.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of Low level laser therapy (LLLT) on stability and displacement of orthodontic miniscrew implants with mediate and immediate force application. They will be assessed 48 miniscrew implants placed in patients in orthodontic treatment at the postgraduate clinical in Orthodontics, at School of Dentistry of Ribeirão Preto, University of São Paulo. They will be randomly divided into 4 groups: 1- LLLT and immediate force application; 2- LLLT and force application 4 weeks after implantation; 3- immediate force application without LLLT and 4- force application 4 weeks after implantation without LLLT. Orthodontic force of 150 gF will be applied for 3 months. A low power laser device Therapy XT with a wavelength of 660 nm and output of 100 mW immediately after implantation (energy density: 4J/cm2), and 808 nm with 100 mW (energy density: 8J/cm2), every 48 hours for two weeks in the following applications will be used. The stability will be assessed using Resonance Frequency Analysis (RFA) at three times: the implantation day (T1), one month (T2) and after 3 months of force application (T3). Stability measures will be evaluated in Implant Stability Quotient (ISQ). To assess the amount of miniscrew implant displacement, it will be used Cone Beam Computed Tomography (CBCT) at the beginning (CT1) and final of the application of orthodontic force (CT2). Three-dimensional models will be created in specific programs and superimpositions of CT1 and CT2 will be used to measure the distance in millimeters between inicial and final position. The evaluation will be carried out in three points: head of miniscrew implant (point C), thread (point R) and apex of miniscrew implant (point A). The results will be statistically analyzed according to nature of the data and the significance level to be adopted will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patient with permanent teeth.
* Use of miniscrews in orthodontic planning.
* Miniscrews placed in the labial upper and lower posterior regions.
* Patient who agree to participate (Informed consent)

Exclusion Criteria:

* Patient with systemic disease.
* Patient with periodontal disease and/or inadequate oral hygiene.
* Use of drugs chronically.
* Patients that consume alcohol or tobacco.
* Use of fixed palatal or lingual orthodontic devices.

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline miniscrew implant stability at 1 and 3 months of force application. | T1: Implantation day; T2: after 1 month; and, T3: after 3 months of force application.
  It will be used a Resonance frequency analysis (RFA) equipment. Stability measures will be evaluated using a unique unit of measure: Implant stability quotient (ISQ). All groups will be evaluated the day of the implantation (T1) and after 1 month (T2).The last stability measure (T3) will be done 3 months after the implantation day in the groups without mediate force application, and 4 months after the implantation day in the groups with mediate force application.
Change from baseline miniscrew implant position at 3 months of force application. | CT1: Implantation day; and, CT2: 3 months of orthodontic force application.
  It will be used Cone Beam Computed tomography (CBCT). Three-dimensional models will be created in specific programs and superimpositions of CT1 and CT2 will be used to measure the distance in millimeters between initial and final position.

CONTACTS AND LOCATIONS:
Overall Officials: Guido A Marañón Vásquez, DDS, Principal Investigator — University of Sao Paulo